CLINICAL TRIAL: NCT03264118
Title: Effects of Antimicrobial Photodynamic Therapy Associated to Biomaterials on Regeneration of Class II Furcation Lesions
Brief Title: Effects of Antimicrobial Photodynamic Therapy on Regeneration of Class II Furcation Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Geistlich Pharma AG (Industry)
Responsible Party: Principal Investigator, Carla Andreotti Damante, Associate professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BauruSchoolDentistryfurcation
Record Dates: First submitted 2017-08-24; First posted 2017-08-28 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Periodontitis, Chronic; Periodontal Diseases; Periodontal Bone Loss
Keywords: Periodontal Guided Tissue Regeneration; Photochemotherapy
MeSH Terms: conditions — Chronic Periodontitis; Periodontal Diseases; Alveolar Bone Loss | interventions — Tooth Exfoliation; Root Planing; Tolonium Chloride

STUDY DESIGN:
Intervention Model Description: Split-mouth design. One side of mouth is test and the other is control side.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Decontamination of furcation defect with scaling and root planing only.
  Interventions: Procedure: Scaling and root planing
- Antimicrobial Photodynamic Therapy (Experimental): Decontamination of furcation defect with scaling and root planing complemented by antimicrobial photodynamic therapy.
  Interventions: Procedure: Scaling and root planing; Drug: Toluidine Blue O

INTERVENTIONS:
Procedure: Scaling and root planing — Furcation treatment by scaling and root planing
Drug: Toluidine Blue O — Antimicrobial photodynamic therapy with toluidine blue O (10mg/ml) and red laser.
  Other Names: Antimicrobial photodynamic therapy
  Arms: Antimicrobial Photodynamic Therapy

SUMMARY:
The aim of this study is to evaluate the additional effect of antimicrobial photodynamic therapy regeneration treatment of mandibular furcation lesions when associated to bovine bone and porcine collagen membrane.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of class II furcation lesion in mandibular 1st and 2nd molars
* Mandibular 1st and 2nd molars without caries, erosion or abrasion

Exclusion Criteria:

* Smoking habit
* Pregnancy
* Use of antibiotics in the last six months
* Periodontal treatment in the last six months
* Endodontic lesion
* Systemic diseases that impair wound healing

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-04-02 (Actual); Primary Completion 2018-12-22 (Actual); Study Completion 2018-12-22 (Actual)

PRIMARY OUTCOMES:
Horizontal probing depth | one year
  Measured with a periodontal probe (mm). Ideal if 0.
Tomographic Bone filling | One year
  Complete filling of furcation defect in tomographic images. Ideal is a radiopaque image similar to neighbor bone.

SECONDARY OUTCOMES:
Probing depth | one year
  Distance from gingival margin to bottom of sulcus. Measured with a periodontal probe (mm). Ideal if < 2 mm.
Clinical Attachment Level | one year
  Distance from cemento-enamel junction to bottom of sulcus. Measured with a periodontal probe (mm). Ideal if < 2 mm.
Bleeding on probing | One year
  Visual confirmation of bleeding after probing. Ideal if not bleeding.

CONTACTS AND LOCATIONS:
Locations (2):
- Brazil (2):
  - Bauru School of Dentistry, Bauru, São Paulo
  - Bauru School of Dentistry, Bauru

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Luchesi VH, Pimentel SP, Kolbe MF, Ribeiro FV, Casarin RC, Nociti FH Jr, Sallum EA, Casati MZ. Photodynamic therapy in the treatment of class II furcation: a randomized controlled clinical trial. J Clin Periodontol. 2013 Aug;40(8):781-8. doi: 10.1111/jcpe.12121. Epub 2013 Jun 3. PMID 23731242
- [Background] Avila-Ortiz G, De Buitrago JG, Reddy MS. Periodontal regeneration - furcation defects: a systematic review from the AAP Regeneration Workshop. J Periodontol. 2015 Feb;86(2 Suppl):S108-30. doi: 10.1902/jop.2015.130677. PMID 25644295